CLINICAL TRIAL: NCT05065463
Title: A Single Dose, Non-randomised, Open-label, Parallel Group Study to Assess the Pharmacokinetics, PCSK9 Reduction, Safety, and Tolerability of AZD8233 in Participants With Severe Renal Impairment, End Stage Renal Disease and Healthy Participants as Controls
Brief Title: To Assess the Pharmacokinetics, Safety, and Tolerability of AZD8233 in Participants With Chronic Kidney Disease (CKD), End Stage Renal Disease (ESRD) and Healthy Participants.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A decision has been taken to discontinue the development of AZD8233 (PCSK9-ASO for sc administration) due to low likelihood of demonstrating a benefit significantly above the current standard of care for patients with high-risk hypercholesterolemia.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7990C00007; 2021-003044-24 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease (ESRD); Renal Impairment; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with severe renal impairment will receive a single dose of AZD8233 on Day 1.
  Interventions: Drug: AZD8233
- Cohort 2 (Experimental): Participants who are healthy will receive a single dose of AZD8233 on Day 1.
  Interventions: Drug: AZD8233
- Cohort 3 (Experimental): Participants with ESRD on dialysis will receive a single dose of AZD8233 on Day 1.
  Interventions: Drug: AZD8233

INTERVENTIONS:
Drug: AZD8233 — Participants will receive a single subcutaneous (SC) dose of AZD8233 into the region of the abdomen.

SUMMARY:
The study is intended to assess the pharmacokinetics (PK), proprotein convertase subtilisin/kexin type 9 (PCSK9) reduction, safety and tolerability of AZD8233 in male and female participants with severe renal impairment and participants with ESRD compared to matched healthy control participants.

DETAILED DESCRIPTION:
This is an open-label, single dose, non-randomised, parallel group study. Participant will be enrolled in 3 cohorts.

* Cohort 1 will include 8 participants with severe renal impairment (estimated glomerular filtration rate [eGFR] of ≥15 to < 30 mL/min/1.73 m^2).
* Cohort 2 will include 8 healthy participants with normal renal function (eGFR of ≥ 90 mL/min/1.73 m^2) that will serve as matched controls for Cohort 1 and Cohort 3. Matching will account for age, Body mass index (BMI), and gender.
* Cohort 3 will include 8 participants with ESRD on dialysis (eGFR of < 15 mL/min/1.73 m^2).

  * Participants in Cohort 3 will receive a single dose of AZD8233 the day after haemodialysis.

Participant will receive the study drug on Day 1, discharged on Day 2 followed by out-patient follow-up visits on Day 3, 7, 14, 28, 42, 56, and 90.

ELIGIBILITY:
Inclusion Criteria:

1. For Cohort 1 and 3 (CKD/ESRD): Participants that are on statins, ACEi/ARB, beta-blocker, diuretic or on any other cardio-renal relevant treatment, the dose should be stable at least 4 weeks prior to Screening (Visit 1) (no dose adjustments within 4 weeks prior to Screening [Visit 1]).
2. For Cohort 2 (HV): Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. (a) Have an eGFR of ≥ 90 mL/min/1.73 m^2 as determined at Screening (Visit 1) via the CKD-EPI formula.
3. For Cohort 1 (CKD): Participants who are severely renally impaired.

   (a) Have an eGFR of ≥15 to < 30 mL/min/1.73 m^2 as determined at Screening (Visit 1) via the CKD-EPI formula.
4. For Cohort 3 (ESRD): Participants with ESRD on dialysis.

   1. Have an eGFR of < 15 mL/min/1.73 m^2.
   2. Have been on stable intermittent haemodialysis for at least 3 months prior to Screening (Visit 1).
5. Body weight of at least 50 kg and BMI within the range ≥ 18 to ≤ 35 kg/m^2 (inclusive).
6. Female of non-childbearing potential or male. Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Participant has a positive SARS-CoV-2 test result within 2 weeks before screening (Visit 1) or between screening and admission to study centre (Day -22 to Day - 2).
2. Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnoea, sore throat, fatigue) 2 weeks before screening (Visit 1) or between screening and admission to study centre (Visit 2).
3. Participant has been previously hospitalised with COVID-19 infection within the last 3 months prior to Screening (Visit 1).
4. Known or suspected history of substance dependence or a positive screen for drugs or alcohol abuse at the Screening Visit.
5. Any laboratory values with the following deviations at the Screening Visit (Visit 1); test may be repeated at the discretion of the Investigator if abnormal:

   (a) Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and HIV. (b) Alanine aminotransferase > 1.5 × ULN (c) Aspartate aminotransferase > 1.5 × ULN (d) Total bilirubin > ULN (e) Haemoglobin < 9 g/dL (f) Platelet count ≤ LLN
6. Previous allogeneic bone marrow transplant.
7. Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

9. Participants with a known hypersensitivity to AZD8233 or any of the excipients of the product.

10. For Cohort 2: Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment,), skin disorder, history of, or ongoing clinically significant allergy/hypersensitivity.

11. Cohort 1 & 3: Presence of unstable medical (e.g., diabetes) or psychological conditions and renal transplant patients.

12. Previous administration of AZD8233/AZD6615 or inclisiran (LEQVIO®, Novartis).

13. Current or previous treatment with drugs for reduction of PCSK9 (for example evolocumab, alirocumab or inclisiran).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | Baseline, 24 hour post-dose, Day 3, 7, 14, 28, 42, 56 and 90
  The pharmacokinetics (PK) parameter of AZD8233 full-length antisense oligonucleotide (ASOs) in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using plasma concentrations. Cmax is defined as observed maximum plasma concentration of AZD8233.
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUCinf) | Baseline, 24 hour post-dose, Day 3, 7, 14, 28, 42, 56 and 90
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using plasma concentrations. AUCinf is defined as area under the plasma concentration-time curve from time zero extrapolated to infinity of AZD8233. AUCinf is estimated by AUClast + Clast/λz where Clast is the observed last quantifiable drug concentration.
Area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUClast) | Baseline, 24 hour post-dose, Day 3, 7, 14, 28, 42, 56 and 90
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using plasma concentrations. AUClast is defined as area under the plasma concentration-curve from time zero to time of last quantifiable concentration of AZD8233.
Area under the concentration-time curve from time zero to 24 hours after dosing (AUC0-24) | Baseline, 24 hour post-dose
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using plasma concentrations. AUC0-24 is defined as area under the concentration-time curve from time zero to 24 hours after dosing of AZD8233.
Renal clearance (CLR) | Post-dose (0-8 hour and 8-24 hour) at Day 1
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using urine concentrations. CLR is defined as renal clearance of AZD8233 from plasma.
Amount excreted in urine (Ae) | Post-dose (0-8 hour and 8-24 hour) at Day 1
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using urine concentrations. The PK urine parameters for AZD8233 full-length ASOs will be derived from Ae. Ae(0-last) is defined as cumulative amount of analyte excreted unchanged in urine at the last sampling interval of AZD8233.
Fraction unbound in plasma (fe) | Post-dose (0-8 hour and 8-24 hour) at Day 1
  The PK of AZD8233 full-length ASOs in participants with severe renal impairment and ESRD compared to matched healthy control participants will be assessed using urine concentrations. The PK urine parameters for AZD8233 full-length ASOs will be derived from fe. fe(0-last) is defined as percentage of dose excreted unchanged in urine from time zero to the last measured time-point for an analyte of AZD8233.
Number of participants with adverse events (AEs) | Day 1 to Day 90
  To assess safety and tolerability of AZD8233 in participants with severe renal impairment, ESRD and their healthy matched controls.

SECONDARY OUTCOMES:
Percentage reduction in proprotein convertase subtilisin/kexin type 9 (PCSK9) plasma levels from baseline | Baseline, 24 hour post-dose, Day 3, 7, 14, 28, 42, 56 and 90
  To asses the percentage change from baseline in PCSK9 plasma levels over-time in participants with severe renal impairment and ESRD compared to their healthy matched controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the requests portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home